CLINICAL TRIAL: NCT05684406
Title: Mitochondrial DNA Copy Number and Leukocyte Telomere Length as Biomarkers in Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Muhammed Naguib Omar, assistant lecturer, Sohag University
Other Study IDs: Soh-Med-22-12-19
Record Dates: First submitted 2022-12-23; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: patients with type 2 diabetes mellitus
  Interventions: Genetic: Genotyping
- Group II: apparently healthy controls with no chronic illness of matched age and sex
  Interventions: Genetic: Genotyping

INTERVENTIONS:
Genetic: Genotyping — Genotyping by Real Time PCR

SUMMARY:
Type 2 diabetes mellitus, which is characterised by a combination of insulin resistance and insufficient insulin secretion is a major contributor to the burden of morbidity and mortality worldwide.

the mitochondrial genome contains multiple copies per cell. Because of its close proximity with higher levels of reactive oxidative species, mitochondrial DNA is prone to oxidative stress; which may lead to mitochondrial dysfunction, characterized by lowered oxidative capacity and reduction in energy production. Mitochondrial dysfunction is associated with aging process and can affect cellular functions and thereby results in a variety of human diseases such as cancer, neurodegenerative diseases, cardiovascular diseases, diabetes and metabolic syndrome .

Telomere length reflects the cumulative damage from those exposure factors and can be used as a potential indicator of biological aging. Shorter telomere length has been linked to the development of a variety of age-related diseases, such as cancer, cardiovascular disease and diabetes

DETAILED DESCRIPTION:
Type 2 diabetes mellitus, which is characterised by a combination of insulin resistance and insufficient insulin secretion is a major contributor to the burden of morbidity and mortality worldwide .The number of adults with type 2 diabetes mellitus is increasing worldwide and if the trend continues the number will rise to 693 million by 2045. Multiple risk factors have been associated with an increased risk of developing type 2 diabetes, including obesity, adverse lifestyle and genetic factors .

Mitochondria generate most of the cell's need for chemical energy in the form of ATP, and mitochondrial dysfunction has been implicated in various aspects of the development and complications of type 2 diabetes including insulin resistance, obesity and beta cell dysfunction. Mitochondrial DNA is a circular and double-stranded DNA molecule comprising 37 genes, of which 13 genes are involved in the electron transport chains and generation of ATP to provide energy for cells, while the remaining genes encode proteins involved in the assembly of amino acids into functional proteins . Unlike the nuclear genome, which normally has only two copies per cell, the mitochondrial genome contains multiple copies per cell. Because of its close proximity with higher levels of reactive oxidative species (ROS), mitochondrial DNA (mtDNA) is prone to oxidative stress; which may lead to mitochondrial dysfunction, characterized by lowered oxidative capacity and reduction in energy production. Mitochondrial dysfunction is associated with aging process and can affect cellular functions and thereby results in a variety of human diseases such as cancer, neurodegenerative diseases, cardiovascular diseases, diabetes and metabolic syndrome.On the other hand, improvement in mitochondrial function, even after critical illness, has been shown to be associated with better survival. Mitochondrial copy number (mtDNA-CN) is a surrogate marker of mitochondrial function . Higher mtDNA-CN is a biomarker of better mitochondrial function and vice versa. A lower mtDNA-CN has been observed in skeletal muscle and adipose tissue of individuals with obesity or type 2 diabetes .similarly, a lower mtDNA-CN in beta cells has also been associated with decreased beta cell function .

In recent years, the association between diabetes mellitus and accelerated biological aging, evaluated by the emerging biomarker (telomere length), has gained much attention.

Telomeres are DNA-protein complexes that cap the chromosomal DNA ends, which preserve genomic integrity and stability. Telomeres shorten during somatic cell division because DNA polymerase is unable to fully replicate the 3' end of DNA. This process can be reversed by an enzyme (telomerase) that is only active in certain replicating tissues, such as male germ cells and activated lymphocytes, stem cells and cancer cells . In normal human cells, telomerase levels are insufficient to maintain telomere length during cell division. When telomeres reach a critically short length, cell growth becomes limited and undergoes cellular senescence or apoptosis. Oxidative stress and chronic inflammation accelerate telomere attribution, resulting in replicative senescence and organ degeneration.Telomere length reflects the cumulative damage from those exposure factors and can be used as a potential indicator of biological aging. Shorter telomere length has been linked to the development of a variety of age-related diseases, such as cancer, cardiovascular disease and diabetes

ELIGIBILITY:
Inclusion Criteria:

* This study will include patients who have type 2 diabetes mellitus.

Exclusion Criteria:

* • Patients who have any other chronic illness.

  * Patients who have cancer.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus aged from 15 years and above, in internal medicine department of Sohag University Hospital and healthy controls of matched age and sex
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
evaluate the potential of peripheral blood mtDNA-CN as biomarker in type 2 diabetic patients | within 3 days after collection of samples
  evaluate the potential of peripheral blood mtDNA-CN as biomarker in type 2 diabeticients pat patients by Real Time PCR

SECONDARY OUTCOMES:
evaluate the potential of leukocyte telomere length as biomarker in type 2 diabetic patients | within 3 days after collection of samples
  evaluate the potential of leukocyte telomere length as biomarker in type 2 diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Hend Muhammed Naguib, Principal Investigator — Sohag University
Locations (1):
- Sohag Univversity, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided